CLINICAL TRIAL: NCT02517528
Title: An Open-Label Study to Evaluate the Safety and Efficacy of ABT-450/Ritonavir/ABT-267 (ABT 450/r/ABT-267) and ABT-333 Coadministered With Ribavirin (RBV) in Treatment-Naïve and Treatment-Experienced Asian Adults With GT1b Chronic Hepatitis C Virus (HCV) Infection and Compensated Cirrhosis
Brief Title: ABT-450/Ritonavir/ ABT-267 (ABT-450/r/ABT-267) and ABT-333 Co-Administered With Ribavirin (RBV) in Treatment Naïve and Treatment Experienced Asian Adults With Genotype 1b Chronic Hepatitis C Virus (HCV) Infection and Compensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-491
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-01

CONDITIONS: Chronic Hepatitis C Virus (HCV)
Keywords: HCV Infection; Compensated Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ombitasvir; paritaprevir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABT-450/r/ABT-267 + ABT-333 + Ribavirin (Experimental): ABT-450/r/ABT-267 once daily + ABT-333 twice daily + weight-based RBV divided twice daily for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267; Drug: ABT-333; Drug: ribavirin

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — Tablet
  Other Names: ombitasvir/paritaprevir/ritonavir; ombitasvir also known as ABT-267; paritaprevir also known as ABT-450
Drug: ABT-333 — Tablet
  Other Names: dasabuvir
Drug: ribavirin — Tablet

SUMMARY:
This is a Phase 3, open-label, multicenter study evaluating the efficacy and safety of ABT-450/r/ ABT-267 and ABT-333 coadministered with RBV for 12 weeks in HCV genotype 1b, treatment naïve and Interferon (IFN) (alpha, beta or pegIFN) plus RBV treatment-experienced Asian adults with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese, South Korean, and Taiwanese descent with full Chinese, South Korean, and Taiwanese parentage.
2. Chronic HCV-infection prior to study enrollment.
3. Screening laboratory result indicating HCV genotype 1b-infection.
4. Compensated cirrhosis defined as a Child-Pugh Score of less than or equal to 6 at Screening.
5. Per local standard practice, documentation of cirrhosis by one of the following methods:

   * Diagnosis on previous liver biopsy or liver biopsy conducted during screening e.g., Metavir Score of > 3 (including 3/4 or 3 - 4), Ishak score of > 4 or,
   * FibroScan score ≥ 14.6 kiloPascals (kPa) within 6 months of Screening or during the Screening Period.

Exclusion Criteria:

1. HCV genotype performed during screening indicating unable to genotype or infection with any other HCV genotype.
2. Positive test result at Screening for Hepatitis B surface antigen (HBsAg), or hepatitis B virus (HBV) DNA > Lower Limit of Quantification (LLOQ) if HBsAg negative, or anti-Human Immunodeficiency virus antibody (HIV Ab).
3. Use of known strong inducers of cytochrome P450 3A (CYP3A) or strong inhibitors of CYP2C8 within 2 weeks or within 10 half-lives, whichever is longer, of the respective medication/supplement prior to study drug administration.
4. Any current or past clinical evidence of Child-Pugh B or C classification or clinical history of liver decompensation including ascites (noted on physical exam), variceal bleeding, or hepatic encephalopathy.
5. Serum Alpha-Fetoprotein (sAFP) > 100 ng/mL at Screening.
6. Confirmed presence of hepatocellular carcinoma (HCC) indicated on imaging techniques such as computed tomography (CT) scan or magnetic resonance imaging (MRI) within 3 months prior to Screening or on an ultrasound performed at Screening (a positive ultrasound result should be confirmed with CT scan or MRI.)
7. Any primary cause of liver disease other than chronic HCV-infection, including but not limited to the following:

   * Hemochromatosis
   * Alpha-1 antitrypsin deficiency
   * Wilson's disease
   * Autoimmune hepatitis
   * Alcoholic liver disease
   * Drug-related liver disease Steatosis and steatohepatitis on a liver biopsy coincident with HCV-related changes would not be considered exclusionary unless the steatohepatitis is considered to be the primary cause of the liver disease.
8. Screening laboratory analyses showing abnormal kidney, hepatic, or hematologic function.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2017-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zha J, Ding B, Wang H, Zhao W, Yu C, Alves K, Mobashery N, Luo Y, Menon RM. Pharmacokinetics of Ombitasvir, Paritaprevir, Ritonavir, and Dasabuvir in Healthy Chinese Subjects and HCV GT1b-Infected Chinese, South Korean and Taiwanese Patients. Eur J Drug Metab Pharmacokinet. 2019 Feb;44(1):43-52. doi: 10.1007/s13318-018-0492-8. PMID 29909549

RESULTS

PARTICIPANT FLOW:
Groups:
- ABT-450/r/ABT-267 + ABT-333 + Ribavirin: ABT-450/r/ABT-267 once daily + ABT-333 twice daily + weight-based ribavirin (RBV) divided twice daily for 12 weeks
Period: Overall Study
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
Started | 104
Completed | 103
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.43 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 40
Region of Enrollment [Number; unit: participants]
  China | 63
  South Korea | 21
  Taiwan | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks Post-Treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ) at 12 weeks following therapy. 95% confidence interval (CI) is calculated using Wilson's score method. The lower bound of the 95% CI for the percentage of participants with SVR12 must exceed 67% to achieve superiority.
Time Frame: 12 weeks after last dose of study drug
Population: Intent-to-Treat Population: all enrolled participants who received at least one dose of study drug. Participants with missing data were imputed as failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
Number analyzed (Participants) | 104
percentage of participants | 100 [96.4 to 100.0]

2. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks Post-Treatment (SVR24)
Description: SVR24 is defined as HCV RNA less than the LLOQ at 24 weeks following therapy. 95% CI is calculated using Wilson's score method. The lower bound of the 95% CI for the percentage of participants with SVR12 must exceed 67% to achieve superiority. SVR24 is primary outcome measure only for China.
Time Frame: 24 weeks after last dose of study drug
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
Number analyzed (Participants) | 104
percentage of participants | 100 [96.4 to 100.0]

3. Secondary Outcome: Percentage of Participants With On Treatment Virologic Failure
Description: On treatment virologic failure is defined as confirmed HCV RNA greater than or equal to the LLOQ at any point during treatment after HCV RNA less than LLOQ, confirmed increase from the lowest value post-baseline in HCV RNA (two consecutive HCV RNA measurements greater than 1 log10 IU/mL above the lowest value post-baseline) at any time point during treatment, or HCV RNA greater than or equal to LLOQ persistently during treatment with at least 6 weeks (greater than or equal to 36 days) of treatment. 95% CI is calculated using Wilson's score method.
Time Frame: Within 12 weeks after first dose of study drug
Population: Intent-to-Treat Population: all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
Number analyzed (Participants) | 104
percentage of participants | 0 [0.0 to 3.6]

4. Secondary Outcome: Percentage of Participants With Virologic Relapse
Description: Virologic relapse is defined as confirmed HCV RNA greater than or equal to LLOQ between end of treatment and 12 weeks after the last dose of study drugs among participants completing treatment and with HCV RNA less than LLOQ at the end of treatment. Completion of treatment is defined as a study drug duration greater than or equal to 77 days. 95% CI is calculated using Wilson's score method.
Time Frame: Within 12 weeks after the last dose of study drug
Population: Intent-to-Treat Population: all enrolled participants who received at least one dose of study drug. Only completers (ie, participants who were dosed with study drug at least 77 days) were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
Number analyzed (Participants) | 103
percentage of participants | 0 [0.0 to 3.6]

5. Secondary Outcome: Percentage of Participants With Virologic Relapse by Post-Treatment Week 24
Description: Virologic relapse is defined as confirmed HCV RNA greater than or equal to LLOQ between end of treatment and 24 weeks after the last dose of study drugs among participants completing treatment and with HCV RNA less than LLOQ at the end of treatment. Completion of treatment is defined as a study drug duration greater than or equal to 77 days. 95% CI is calculated using Wilson's score method.
Time Frame: Within 24 weeks after the last dose of study drug
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
Number analyzed (Participants) | 103
percentage of participants | 0 [0.0 to 3.6]

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs) collected from Screening through Post-Treatment Week 48 (or discontinuation); AEs collected from Screening through 30 days post-dosing.
Arm/Group | ABT-450/r/ABT-267 + ABT-333 + Ribavirin
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 4/104
Other Adverse Events (participants affected / at risk) | 71/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-450/r/ABT-267 + ABT-333 + Ribavirin (N=104)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1)
FOOD POISONING (Gastrointestinal disorders) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1)
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-450/r/ABT-267 + ABT-333 + Ribavirin (N=104)
ANAEMIA (Blood and lymphatic system disorders) | 15 (15)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (7)
ASTHENIA (General disorders) | 12 (13)
FATIGUE (General disorders) | 11 (11)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 12 (12)
BLOOD BILIRUBIN INCREASED (Investigations) | 26 (27)
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 12 (14)
HAEMOGLOBIN DECREASED (Investigations) | 7 (10)
RETICULOCYTE COUNT INCREASED (Investigations) | 6 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 (8)
DIZZINESS (Nervous system disorders) | 11 (15)
HEADACHE (Nervous system disorders) | 7 (12)
INSOMNIA (Psychiatric disorders) | 6 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (14)
PRURITUS (Skin and subcutaneous tissue disorders) | 16 (18)
RASH (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-02-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT02517528/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02517528/SAP_001.pdf